CLINICAL TRIAL: NCT03074344
Title: Study on the Effectiveness of Eye-drops Containing Cross-linked Hyaluronic Acid and Coenzyme Q10 in the Treatment of Patients With Mild to Moderate Dry Eye
Brief Title: Cross-linked Hyaluronic Acid and Coenzyme Q10 in the Treatment of Dry Eye
Acronym: DEDCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Policlinico "G. Martino" (Other)
Responsible Party: Principal Investigator, Pasquale Aragona, Full Professor of Ophtalmology, Azienda Ospedaliera Universitaria Policlinico "G. Martino"
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AOUGMartino
Record Dates: First submitted 2017-02-28; First posted 2017-03-08 (Actual); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Dry Eye Syndrome
Keywords: Dry Eye Syndrome; artificial tear; CoQ10; Hyaluronic acid
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Randomised, single-masked, parallel-group comparative study.
Who Masked: Investigator
Masking Description: Visits were carried out in a blind fashion by investigators who were not aware to which group the patients belonged. The patients were allowed to know the brand name of the eye drops they were using.
Oversight: Data Monitoring Committee: No

ARMS (2):
- XLHA+CoQ10 (Experimental): XLHA+CoQ10 eye drop administered four times a day for 12 weeks (90 days).
  Interventions: Device: XLHA+CoQ10
- Hyaluronic acid (HA) (Active Comparator): Hyaluronic acid (HA) eye drop administered four times a day for 12 weeks (90 days).
  Interventions: Device: Hyaluronic acid (HA)

INTERVENTIONS:
Device: XLHA+CoQ10 — XLHA+CoQ10 for four times a day for 12 weeks.
  Other Names: VisuXL®
  Arms: XLHA+CoQ10
Device: Hyaluronic acid (HA) — Hyaluronic acid (HA) for four times a day for 12 weeks.
  Arms: Hyaluronic acid (HA)

SUMMARY:
Background: Dry eye disease (DED) is a common condition causing burden on visual function and reducing quality of life. Corticosteroids and/or cyclosporine eye drops are able to improve DED symptoms, however, side effects of immune suppression and cost lead patients often to suspend treatment. Consequently, is important to identify therapies alleviating DED symptoms. A randomized, controlled, single masked study, was performed in 40 patients affected by mild to moderate DED, to evaluate efficacy and safety of a collyrium based on cross-linked hyaluronic acid (XLHA) added with Coenzyme Q10 (CoQ10) in comparison to an eye drop considered a gold standard for tear substitutes, based on hyaluronic acid (HA) 0.15%.

Methods: eye drops were administered four times a day for 90 days to enrolled subjects divided in two groups: group A treated with XLHA+CoQ10, group B treated with HA. Ocular Surface Disease Index (OSDI) questionnaire, visual acuity, intraocular pressure (IOP), fundus exam, tear break-up time (TBUT), corneal and conjunctival fluorescein staining, corneal esthesiometry, corneal confocal microscopy, were performed at different visits until the 90th day.

DETAILED DESCRIPTION:
Introduction:

Dry eye disease (DED) is a common eye condition causing burden on visual function and reducing quality of life and work productivity. DED is a tear film disorder resulting in hyperosmolarity of tear film and inflammation of ocular surface that results in symptoms of discomfort, visual disturbance, and tear film instability with potential damage to the ocular surface. This condition provokes traumatisms caused by the movement of the eyelids on the ocular surface and an insufficient cleansing of the same by microbial agents and/or foreign bodies.

Prevalence of DED increases with age and women are particularly susceptible, especially those receiving estrogens. The pathogenesis is not fully understood; however, it has been recognized that inflammation has a prominent role .

The most common symptoms of DED are: burning, foreign body sensation in the eye, difficulty in opening the eyelids on awakening, blurred vision and, in severe cases, pain and photophobia. DED is accompanied by increased tear film osmolarity and inflammation of ocular surface.

There is no gold standard treatment for DED, but corticosteroids and/or cyclosporine eye drops improve the symptoms. However, given the side effects of immune suppression and the cost of pharmaceutical preparations, patients often suspend treatment before the effectiveness of therapy can be verified.

Artificial tears are considered a mainstay in dry eye treatment. Hyaluronic acid (HA), a natural glycosaminoglycan, is a component of tear film. It increases tear film viscosity and hydrates and lubricates the ocular surface. HA possesses intrinsic water retention properties, viscoelasticity and favours the healing of corneal and conjunctival epithelium. Safety and efficacy of HA for the treatment of DED has been demonstrated. Eye-drops containing HA determine a reduction of ocular surface inflammation, with consequent improvement of quality of corneal and conjunctival epithelium. Our previous clinical study showed HA beneficial effects on the conjunctival epithelium of dry eye patients. Results of another clinical trial, confirm beneficial effects of HA and show that in combination with tamarind seed polysaccharide it can be effective in improving dry eye symptoms, opening new scenarios in the treatment of this disease by combining different molecules.

Coenzyme Q10 (CoQ10) is an endogenous, lipid soluble molecule, also known as ubiquinone. CoQ10 plays a key role in oxidative metabolism supporting the adenosine triphosphate (ATP) in the mitochondria and, in its reduced form, acts as a lipid antioxidant. In almost all tissues of the human body, CoQ10 levels decline with age and ocular function is sensitive to variations of concentration of CoQ10 .

A randomized, controlled, single masked study, was performed in mild to moderate dry eye patients, to evaluate the efficacy and the safety of a collyrium based on cross-linked HA (XLHA) added with CoQ10 in comparison to an eye drop formulation, commonly used in clinical practice and considered a gold standard for tear substitutes, in the treatment of dry eye, based on 0.15% linear HA.

Methods This randomised, single-masked, parallel-group comparative study investigated the efficacy and safety, in treatment of dry eye patients, of an ophthalmic solution containing XLHA added with CoQ10 (VisuXL®, Visufarma, Rome, Italy) in comparison with a formulation containing hyaluronic acid 0.15% (HA). The study screened 46 patients and 40 were enrolled [(13 male, 17 female, with an age range 40-79 years; mean age 62 ± 12.8 (SD) years)] suffering from mild to moderate dry eye attending to the Eye Clinic, Department of Biomedical Sciences, Regional Referral Center for the Ocular Surface Diseases, University of Messina, Messina, Italy. Enrolled subjects were divided into two treatment groups (Group A receiving the study formulation based on XLHA+CoQ10 and Group B receiving the comparator formulation based on 0.15% HA) according to a randomization scheme, corresponding to allocation codes generated for the two treatments using the permuted block method. The two eye-drops compositions used for the study were the following: group A formulation (XLHA+CoQ10): 100 ml containing Cross-Linked HA sodium salt 100 mg, Coenzyme Q10 100 mg, with Vitamin E tocopheryl polyethylene glycol succinate (TPGS) 500 mg (as a solubilizing agent for the lipid soluble CoQ10), Isotonic buffered solution q.s. to 100 ml; group B formulation: HA sodium salt 100 mg; isotonic buffered solution q.s. to 100 ml. Both formulations were unpreserved.

All patients included were treated for a run-in period of 7 days with one eye drop of saline four times daily. At the end of this period (time 0 of the study) the subjects were randomly divided into the two groups and assigned to a treatment.

The visits were carried out in a blind fashion by investigators. Eye drops were administered four times a day for 12 weeks and subjects enrolled in the study underwent grading of subjective symptoms and clinical examination at time 0 and after 15, 30, and 90 days. The patients were allowed to know the brand name of the eye drops they were using.

Outcomes The Ocular Surface Disease Index (OSDI) questionnaire, visual acuity, intraocular pressure (IOP), and fundus exam, tear break-up time (TBUT), corneal and conjunctival fluorescein staining, esthesiometry, corneal confocal microscopy. Adverse events were monitored.

OSDI is one of the most widely used questionnaires. The 12-item OSDI questionnaire scores range from 0 to 100, high scores represent higher disability. The scale showed good sensitivity in discriminating normal people from subjects affected by dry eye and to correlate well with disease severity.

The ocular surface fluorescein stain score was assessed 3 minutes after the instillation of fluorescein; a modified Oxford score was used: cornea and conjunctiva were scored separately from 0 to 5 (from 0 = none to 5 = extended areas of confluent stain), for the conjunctiva a mean for the scores from the nasal and temporal regions was used. The ocular surface was observed through a cobalt blue light and a Wratten #12 yellow filter.The difference among the scores obtained in each visit was calculated.

Corneal sensitivity was measured by Cochet-Bonnet aesthesiometer to evaluate the activity of the ophthalmic branch of fifth cranial nerve (trigeminal). It was measured by the evaluating the length of the filament able to evoke a tactile sensation (mm of filament).

In vivo confocal microscopy was performed, after the topical instillation of a drop of unpreserved 0.4% oxybuprocaine, using the 40x contact objective and the additional Z-Ring probe, to allow a precise positioning of the probe over the central corneal area.

For statistical analysis, only the results of right eyes were considered. Student's t-test and Mann-Whitney U-test were used as appropriate. Values of P≤0.05 were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80 years,
* history of at least 3 months of dry eye symptoms referable to mild to moderate dry eye.

Exclusion Criteria:

* presence of any ocular disease, present or past, other than dry eye;
* previous ocular surgery,
* use of contact lens or topic treatments other than tear substitutes;
* presence of systemic diseases requiring a treatment with systemic drugs potentially interfering with tear productions;
* hypersensitivity to the active substance or to excipients;
* participation in a clinical trial during the 3 months prior to the beginning of the study,
* pregnancy or breast-feeding.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-05; Primary Completion 2016-07 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Ocular Surface Disease Index (OSDI) questionnaire. | Up to 90 days.
  The OSDI is assessed on a scale of 0 to 100, with higher scores representing greater disability. OSDI is a valid and reliable instrument for measuring dry eye disease (normal, mild to moderate, and severe) and effect on vision-related function. OSDI demonstrates sensitivity and specificity in distinguishing between normal subjects and patients with dry eye disease.
Corneal and conjunctival staining. | Up to 90 days.
  Corneal and conjunctival staining of the ocular surface after instillation of vital dyes was developed to quantify epithelial surface damage in dry eye patients. Ocular surface fluorescein stain score was assessed 3 minutes after the instillation of fluorescein; a modified Oxford score was used: cornea and conjunctiva were scored separately from 0 to 5 (from 0 = none to 5 = extended areas of confluent stain), for the conjunctiva a mean for the scores from the nasal and temporal regions was used. The ocular surface was observed through a cobalt blue light and a Wratten #12 yellow filter.The difference among the scores obtained in each visit was calculated.

SECONDARY OUTCOMES:
Visual acuity, | Up to 90 days.
  Visual acuity refers to the ability to discern fine distinctions in the environment.
Intraocular pressure (IOP). | Up to 90 days.
  IOP = eye fluid pressure measured by tonometry.
Fundus exam. | Up to 90 days.
  Fundus exam is observed after use of mydriatic drops enlarging the pupil.
Tear break-up time (TBUT). | Up to 90 days.
  Tear breakup time (TBUT) is a test used to assess for evaporative dry eye disease. To measure TBUT, fluorescein is instilled into the patient's tear film then and the patient is asked not to blink while the tear film is observed under cobalt blue illumination. TBUT is recorded as the number of seconds that elapse between the last blink and the appearance of the first dry spot in the tear film, as seen in this progression of these slit lamps photos over time. A TBUT under 10 seconds is considered abnormal.
Corneal esthesiometry. | Up to 90 days.
  Esthesiometry measures sensation, specifically tactile.

CONTACTS AND LOCATIONS:
Overall Officials: Pasquale Aragona, MD, Principal Investigator — Azienda Ospedaliera Universitaria Policlinico "G. Martino", Messina, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benitez-Del-Castillo J, Labetoulle M, Baudouin C, Rolando M, Akova YA, Aragona P, Geerling G, Merayo-Lloves J, Messmer EM, Boboridis K. Visual acuity and quality of life in dry eye disease: Proceedings of the OCEAN group meeting. Ocul Surf. 2017 Apr;15(2):169-178. doi: 10.1016/j.jtos.2016.11.003. Epub 2016 Nov 30. PMID 27913232
- [Background] Al-Saedi Z, Zimmerman A, Bachu RD, Dey S, Shah Z, Baugh R, Boddu SH. Dry Eye Disease: Present Challenges in the Management and Future Trends. Curr Pharm Des. 2016;22(28):4470-90. doi: 10.2174/1381612822666160614012634. PMID 27296759
- [Background] Milner MS, Beckman KA, Luchs JI, Allen QB, Awdeh RM, Berdahl J, Boland TS, Buznego C, Gira JP, Goldberg DF, Goldman D, Goyal RK, Jackson MA, Katz J, Kim T, Majmudar PA, Malhotra RP, McDonald MB, Rajpal RK, Raviv T, Rowen S, Shamie N, Solomon JD, Stonecipher K, Tauber S, Trattler W, Walter KA, Waring GO 4th, Weinstock RJ, Wiley WF, Yeu E. Dysfunctional tear syndrome: dry eye disease and associated tear film disorders - new strategies for diagnosis and treatment. Curr Opin Ophthalmol. 2017 Jan;27 Suppl 1(Suppl 1):3-47. doi: 10.1097/01.icu.0000512373.81749.b7. PMID 28099212
- [Background] The management of dry eye. Drug Ther Bull. 2016 Jan;54(1):9-12. doi: 10.1136/dtb.2016.1.0378. PMID 26763598
- [Background] Schaumberg DA, Sullivan DA, Buring JE, Dana MR. Prevalence of dry eye syndrome among US women. Am J Ophthalmol. 2003 Aug;136(2):318-26. doi: 10.1016/s0002-9394(03)00218-6. PMID 12888056
- [Background] Stevenson W, Chauhan SK, Dana R. Dry eye disease: an immune-mediated ocular surface disorder. Arch Ophthalmol. 2012 Jan;130(1):90-100. doi: 10.1001/archophthalmol.2011.364. PMID 22232476
- [Background] The definition and classification of dry eye disease: report of the Definition and Classification Subcommittee of the International Dry Eye WorkShop (2007). Ocul Surf. 2007 Apr;5(2):75-92. doi: 10.1016/s1542-0124(12)70081-2. PMID 17508116
- [Background] Baudouin C, Aragona P, Van Setten G, Rolando M, Irkec M, Benitez del Castillo J, Geerling G, Labetoulle M, Bonini S; ODISSEY European Consensus Group members. Diagnosing the severity of dry eye: a clear and practical algorithm. Br J Ophthalmol. 2014 Sep;98(9):1168-76. doi: 10.1136/bjophthalmol-2013-304619. Epub 2014 Mar 13. PMID 24627252
- [Background] She Y, Li J, Xiao B, Lu H, Liu H, Simmons PA, Vehige JG, Chen W. Evaluation of a Novel Artificial Tear in the Prevention and Treatment of Dry Eye in an Animal Model. J Ocul Pharmacol Ther. 2015 Nov;31(9):525-30. doi: 10.1089/jop.2015.0042. Epub 2015 Aug 31. PMID 26322539
- [Background] Stocker R, Bowry VW, Frei B. Ubiquinol-10 protects human low density lipoprotein more efficiently against lipid peroxidation than does alpha-tocopherol. Proc Natl Acad Sci U S A. 1991 Mar 1;88(5):1646-50. doi: 10.1073/pnas.88.5.1646. PMID 2000375
- [Background] Fernandez MM, Afshari NA. Nutrition and the prevention of cataracts. Curr Opin Ophthalmol. 2008 Jan;19(1):66-70. doi: 10.1097/ICU.0b013e3282f2d7b6. PMID 18090901
- [Background] Schiffman RM, Christianson MD, Jacobsen G, Hirsch JD, Reis BL. Reliability and validity of the Ocular Surface Disease Index. Arch Ophthalmol. 2000 May;118(5):615-21. doi: 10.1001/archopht.118.5.615. PMID 10815152
- [Background] Sullivan BD, Whitmer D, Nichols KK, Tomlinson A, Foulks GN, Geerling G, Pepose JS, Kosheleff V, Porreco A, Lemp MA. An objective approach to dry eye disease severity. Invest Ophthalmol Vis Sci. 2010 Dec;51(12):6125-30. doi: 10.1167/iovs.10-5390. Epub 2010 Jul 14. PMID 20631232
- [Background] Mandell RB. Slit lamp classification system. J Am Optom Assoc. 1987 Mar;58(3):198-201. PMID 3571821
- [Background] Faulkner WJ, Varley GA. Corneal diagnostic techniques. In: Krachmer JH, Mannis MJ, Holland EJ, eds. Cornea. 2nd ed. Vol. 1 Philadelphia: Elsevier/Mosby; 2005:229-235.
- [Background] Fabiani C, Barabino S, Rashid S, Dana MR. Corneal epithelial proliferation and thickness in a mouse model of dry eye. Exp Eye Res. 2009 Aug;89(2):166-71. doi: 10.1016/j.exer.2009.03.003. Epub 2009 Mar 17. PMID 19298814
- [Result] Aragona P, Papa V, Micali A, Santocono M, Milazzo G. Long term treatment with sodium hyaluronate-containing artificial tears reduces ocular surface damage in patients with dry eye. Br J Ophthalmol. 2002 Feb;86(2):181-4. doi: 10.1136/bjo.86.2.181. PMID 11815344
- [Result] Barabino S, Rolando M, Nardi M, Bonini S, Aragona P, Traverso CE. The effect of an artificial tear combining hyaluronic acid and tamarind seeds polysaccharide in patients with moderate dry eye syndrome: a new treatment for dry eye. Eur J Ophthalmol. 2014 Mar-Apr;24(2):173-8. doi: 10.5301/ejo.5000355. Epub 2013 Sep 9. PMID 24030535
- [Result] Frei B, Kim MC, Ames BN. Ubiquinol-10 is an effective lipid-soluble antioxidant at physiological concentrations. Proc Natl Acad Sci U S A. 1990 Jun;87(12):4879-83. doi: 10.1073/pnas.87.12.4879. PMID 2352956